CLINICAL TRIAL: NCT00030108
Title: Phase I Trial and Pharmacokinetic Study of BMS-247550 (NSC 710428, Ixabepilone), an Epothilone B Analog, in Pediatric Patients With Refractory Solid Tumors and Leukemias
Brief Title: Ixabepilone in Treating Young Patients With Solid Tumors or Leukemia That Haven't Responded to Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 020031; 02-C-0031; NCI-5425; CDR0000069133; NCT00025961 (obsolete NCT alias)
Record Dates: First submitted 2002-01-30; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Kidney Cancer; Leukemia; Liver Cancer; Neuroblastoma; Ovarian Cancer; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood rhabdomyosarcoma; childhood craniopharyngioma; recurrent neuroblastoma; recurrent childhood liver cancer; recurrent Wilms tumor and other childhood kidney tumors; childhood central nervous system germ cell tumor; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific; childhood germ cell tumor; recurrent childhood soft tissue sarcoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor; B-cell childhood acute lymphoblastic leukemia; childhood acute basophilic leukemia; childhood acute eosinophilic leukemia; childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; childhood acute promyelocytic leukemia (M3); L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; L3 childhood acute lymphoblastic leukemia; non-T, non-B, cALLa negative childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive childhood acute lymphoblastic leukemia; non-T, non-B, cALLa positive, pre-B childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; TdT negative childhood acute lymphoblastic leukemia; TdT positive childhood acute lymphoblastic leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Wilms Tumor; Osteosarcoma; Oligodendroglioma; Choroid Plexus Neoplasms; Astrocytoma; Medulloblastoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer; Leukemia, Eosinophilic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of ixabepilone in treating young patients with relapsed or refractory solid tumors or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of ixabepilone in young patients with refractory solid tumors (closed to accrual as of 10/4/2007) or relapsed or refractory leukemia.
* Determine the toxicity spectrum of this drug in these patients.
* Determine the plasma pharmacokinetics of this drug in these patients.
* Determine the pharmacodynamics of this drug in these patients.
* Assess the nerve growth factor levels, before and after the initiation of this drug, as a potential surrogate marker for the development of peripheral neuropathy in these patients.

Secondary

* Determine the response of patients treated with this drug.
* Compare the tolerability, toxicity profile, MTD, DLT, pharmacokinetics, and pharmacodynamics of this drug in young patients treated on this study vs adults with solid tumors (closed to accrual as of 10/4/2007) treated on the ongoing Medicine Branch, NCI, phase I study.
* Assess the safety and tolerability of ixabepilone at the solid tumor MTD (expanded leukemia cohort).
* Evaluate the plasma pharmacokinetics of in young patients with refractory or relapsed leukemia.
* Evaluate the extent of tubulin polymerization in leukemic blasts at baseline after treatment with ixabepilone ex-vivo.
* Compare the effects of tubulin polymerization in leukemic blasts with ixabepilone versus paclitaxel ex-vivo with an without the presence of a potent P-glycoprotein inhibitor.
* Evaluate the activity known drug transporters in drug-resistant leukemias in leukemic blasts.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive ixabepilone IV over 1 hour on days 1-5. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity. Intrapatient dose escalation to one dose level above the enrollment dose level is allowed in patients who have stable or responding disease or are experiencing other benefits from therapy (e.g., decrease in tumor-related pain symptoms) and who have no grade 2 or greater non-hematologic toxicity and no grade 3 or greater hematologic toxicity. Additional patients are treated at the MTD. Patients treated at the MTD may not undergo intrapatient dose escalation.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed solid tumor (closed to accrual as of 10/4/2007) that relapsed after or failed to respond to front-line curative therapy and for which no other potentially curative treatment options exist

    * Curative therapy may include surgery, radiotherapy, chemotherapy, or any combination of these modalities
    * Eligible tumor types include, but are not limited to, the following:

      * Rhabdomyosarcoma
      * Other soft tissue sarcomas
      * Ewing's sarcoma family of tumors
      * Osteosarcoma
      * Neuroblastoma
      * Wilms' tumor
      * Hepatic tumors
      * Germ cell tumors
      * Primary brain tumors

        * Histologic confirmation may be waived for brain stem or optic glioma
  * Diagnosis of relapsed or refractory leukemia

    * Patients with refractory or second or greater relapsed leukemia must have > 25% blasts in the bone marrow (M3 bone marrow) with or without active extramedullary disease (except for leptomeningeal disease)
    * Relapsed after or failed to respond to frontline curative therapy and no other potentially curative therapy (e.g., radiotherapy, chemotherapy, or any combination of these modalities) exists
  * Patients with acute promyelocytic leukemia must be refractory to treatment with retinoic acid and arsenic trioxide
  * Patients with Philadelphia chromosome positive chronic myelogenous leukemia must be refractory to imatinib
* No active CNS leukemia (CNS3)

PATIENT CHARACTERISTICS:

Age:

* 2 to 18 (solid tumor patients [closed to accrual as of 10/4/2007])
* 1 to 21 (leukemia patients)

Performance status:

* For patients age 11 to 21:

  * Karnofsky 50-100%
* For patients age 1 to 10:

  * Lansky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3 (20,000/mm^3 for leukemia patients)
* Hemoglobin ≥ 8.0 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT less than 2.5 times ULN
* No hepatic dysfunction that would preclude study

Renal:

* Creatinine normal for age OR
* Creatinine clearance at least 60 mL/min
* No renal dysfunction that would preclude study

Other:

* No known severe prior hypersensitivity reaction to agents containing Cremophor EL
* No clinically significant unrelated systemic illness (e.g., serious infections or other organ dysfunction) that would preclude study
* No grade 2 or greater preexisting sensory neuropathy
* More than 2 month since prior and no concurrent evidence of graft vs host disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from all therapy-related acute toxic effects (leukemia patients only)
* Prior epoetin alfa allowed
* At least 3 days since other prior colony-stimulating factors (e.g., filgrastim (G-CSF), sargramostim (GM-CSF), or interleukin-11 (IL-11))
* At least 6 months since prior bone marrow transplantation
* At least 2 months since prior stem cell transplantation or rescue (leukemia patients)
* At least 7 days since prior therapy with a biological agent and hematopoietic growth factor with the exception of erythropoietin
* More than 3 weeks since prior monoclonal antibody therapy (leukemia patients only)
* No concurrent GM-CSF or IL-11
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* Recovered from all therapy-related acute toxic effects (leukemia patients only)
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed for the control of symptoms related to tumor-associated edema in patients with brain tumors
* Patients with brain tumors must be on a stable or tapering dose of corticosteroids for 7 days before baseline scan is performed for the purpose of assessing response to study therapy
* Must be on a stable or tapering dose of corticosteroids for 7 days prior to study entry (leukemia patients only)

Radiotherapy:

* See Disease Characteristics
* Recovered from all therapy-related acute toxic effects (leukemia patients only)
* At least 4 weeks since prior radiotherapy
* More than 2 weeks since prior local palliative radiotherapy (leukemia patients only)
* More than 3 months since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥50% of the pelvis (leukemia patients only)
* More than 6 weeks since prior other substantial bone marrow radiotherapy (leukemia patients only)
* No prior extensive radiotherapy (e.g., craniospinal irradiation, total body irradiation, or radiotherapy to more than half of the pelvis)
* No concurrent anticancer radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* At least 30 days since any prior investigational anticancer therapy
* At least 1 week since prior known inhibitors of CYP3A4, including any of the following:

  * Antibiotics (i.e., clarithromycin, erythromycin, or troleandomycin)
  * Anti-HIV agents (i.e, delaviridine, nelfinavir, amprenavir, ritonavir, idinavir, saquinavir, or lopinavir)
  * Anti-fungals (i.e., itraconazole, ketoconazole, fluconazole [doses > 3mg/kg/day], or voriconazole)
  * Anti-depressants (i.e., nefaxodone or fluovoxamine)
  * Calcium channel blockers (i.e., verapamil or diltiazem)
  * Anti-emetics (i.e., aprepitant [Emend®])
  * Miscellaneous agents (i.e., amiodarone)
  * Grapefruit juice
* No other concurrent investigational agents
* No concurrent St. John's Wort
* No concurrent known inhibitors of CYP3A4, including grapefruit juice
* Concurrent other agents inducing CYP3A4 allowed

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-11; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicity of ixabepilone
Toxicity spectrum
Plasma pharmacokinetics
Pharmacodynamics
Nerve growth factor levels before and after drug administration

SECONDARY OUTCOMES:
Objective tumor response
Tubulin polymerization in PBMCs prior to the start of the infusion, just before the end of the infusion, 5 hours after the end of the infusion and before the start of the infusion on day 2 of the ixabepilone on course 1

CONTACTS AND LOCATIONS:
Overall Officials: AeRang Kim, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland

REFERENCES:
- [Result] Widemann BC, Goodspeed W, Goodwin A, Fojo T, Balis FM, Fox E. Phase I trial and pharmacokinetic study of ixabepilone administered daily for 5 days in children and adolescents with refractory solid tumors. J Clin Oncol. 2009 Feb 1;27(4):550-6. doi: 10.1200/JCO.2008.17.6644. Epub 2008 Dec 15. PMID 19075272